CLINICAL TRIAL: NCT05860920
Title: Clinical Diagnostic Performance Evaluation of an Anti-Measles IgM Lateral Flow Immunochromatographic Assay for Outbreak Detection and Surveillance in Senegal
Brief Title: Clinical Diagnostic Performance Evaluation of a Measles Rapid Test in Senegal
Status: Not yet recruiting | Type: Observational
Sponsor: Institut Pasteur de Dakar (Other)
Collaborators: Ministry of Health, Senegal (Other Government); Epicentre (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-01
Record Dates: First submitted 2023-05-03; First posted 2023-05-16 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Measles
MeSH Terms: conditions — Measles

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this study is to measure the accuracy of a new measles rapid test when used in clinical health centres in several regions of Senegal. The rapid test will be used to test patients for measles who attend the participating health centres with signs and symptoms suggestive of measles infection. The rapid test can be used with a drop of blood from a finger, or oral fluid sampled with a swab rubbed over the gums. The rapid test will be compared to the standard methods of diagnosis in the laboratory using blood samples and oral or throat samples taken for surveillance purposes.

The main questions the study aims to answer are:

1. What is the accuracy of the rapid test when used with capillary blood (a drop of blood from the finger tip) in health centres by non-laboratory health professionals?
2. What is the accuracy of the rapid test when used with oral fluid by non-laboratory health professionals?

In addition to measuring the accuracy of the test, data will also be collected on whether the test is easy and practical to use and how best to record the results.

DETAILED DESCRIPTION:
A. Product undergoing evaluation

Anti-measles IgM lateral flow immunochromatographic assay manufactured by DIATROPIX (Dakar, Senegal). The rapid diagnostic test (RDT) will be prepared in kits for use with serum and capillary fluid, with additional devices available for experimental use with oral fluid.

B. Study design

This is a prospective diagnostic evaluation study of a professional use measles RDT, designed to assess the performance (sensitivity and specificity) of the RDT for measles case confirmation by non-laboratory personnel for the purposes of outbreak detection and national surveillance. The RDT performance using capillary blood and oral fluid will be compared to the combined reference standard of detection of anti-measles IgM by ELISA in the serum of a suspected case or a positive PCR result for measles (on nasopharyngeal swab sample or oral fluid). Given that serum samples will be collected for reference testing (as part of usual surveillance practice), the study design will also incorporate an evaluation of the use of the RDT by laboratory staff on serum.

C. Sample size

Using a simulation approach based on 10,000 results we estimate that a minimum of 672 measles IgM-negative and 172 IgM-(or PCR) positive cases (by reference test results) are required to ensure sufficient precision of the sensitivity and specificity estimates to meet Target Product Profile requirements; with a total target sample size of at least 844 depending on the % positivity of tested samples.

D. Recruitment

Recruitment will align with the case-based measles surveillance strategy, whereby consecutive eligible patients that present to the study site will be invited to participate in surveillance. All measles suspected cases will be eligible for testing in line with the national case-based surveillance approach (including those who are epidemiologically linked clinical cases).

Patients meeting the study inclusion criteria will be provided with information concerning the study and the additional diagnostic testing involved beyond what is required for clinical care or routine surveillance. Inclusion will follow an informed consent procedure and individuals who do not wish to participate, will continue to receive routine clinical care, which may include routine surveillance activities.

Urgent clinical care, intervention or referral/transfer to another site will not be delayed, and patients are only eligible for inclusion once clinically stable as deemed by the responsible clinical officer.

E. Clinical sampling strategy

All participants will undergo venous, capillary blood and oral fluid sampling (unless specific exclusions apply). The venous blood draw is aligned to the ministry of health standard operating procedure for surveillance. For the purposes of the study, oral fluid sampling will replace naso-pharyngeal swabbing as an equivalent technique for measles RNA detection.

Venous blood/serum sampling

Venous whole blood will be taken in a plain, dry tube from patients of all ages (unless it is current practice to obtain serum samples using heelstick capillary sampling in young infants at the study site). The whole blood sample will be stored or centrifuged to facilitate serum separation at the participating site in preparation for transport and testing the serum for measles IgM at an Institut Pasteur de Dakar (IPD) laboratory, using both the RDT (10 microlitres) and ELISA (100 microlitres). These sera may also undergo additional testing as part of routine of surveillance, including for rubella and zika IgM.

Oral fluid sampling

Unless ineligible (see oral fluid exclusion criteria) an oral fluid sample will be taken from all participants and added to virus transport medium (VTM)/buffer, as per manufacturer's instructions. Following sample preparation, the oral fluid will be tested on-site for the presence of IgM using the RDT. The residual liquid sample will be stored and transported to the measles national reference laboratory for PCR +/- other molecular testing.

As well as assessing the RDT performance with oral fluid, the collection of this sample alongside serum strengthens the reference standard against which the new RDT is evaluated. It will also allow assessment of the added value of molecular analysis of circulating measles strains to inform national surveillance and guide public health decisions. Therefore, if the participant is ineligible for oral fluid sampling but a nasopharyngeal swab is feasible, this will be taken instead. However, nasopharyngeal swabs samples will not be applied to the RDT.

Capillary blood

All participants will have a capillary blood sample taken using the World Health Organisation (WHO) recommended technique. Capillary blood (5 microlitres) will be added directly to sample buffer as per the standard operating procedure/manufacturer's instructions and following dilution, applied to an RDT without delay. After confirming a valid result on the RDT, the residual diluted capillary blood will be discarded.

F. Rapid diagnostic testing

For each rapid test (serum, capillary blood, oral fluid), the results will be read and interpreted as positive or negative by two independent laboratory staff (for serum) or non-laboratory staff (for capillary blood and oral fluid). Both the qualitative interpretation and the intensity of the control and test lines according to a reference card will be documented, along with the timing of the reading.

Following the reading of the result, a photograph will be taken and the RDT used with capillary blood or oral fluid will be dried, stored with desiccant and transported to IPD for additional molecular analyses.

Staff will receive training on the use of the RDT during study implementation and will be provided with the protocol and product information/manufacturers' instructions for use.

This information will include storage temperature, kit contents, operating temperature, minimum and maximum incubation time, stability of the products after opening, additional equipment or consumables required but not provided in the kit, and number of steps in the procedure.

G. Inter-reader variability

All the RDTs performed will be read by a second investigator and the results will be compared to assess inter-reader variability. Any discrepancies will be resolved by a third independent reading by a trained study team member. The name of the staff member recording each RDT result will be documented. The study team at each participating site/laboratory will be trained to ensure each reading is undertaken independently. The RDT will be performed and interpreted before the ELISA result is known.

H. Study duration

The study will last for the time necessary to include the estimated required sample size (minimum number of positives and negative suspected cases), with a target for completion within 6 months, and the possibility to extend to 9 months. Personnel at the virology reference testing laboratory at IPD, who will be blinded to the RDT results, will monitor the number of positive and negative cases (as per reference testing) every week. The study team will review the overall recruitment progress on a weekly basis, with input from the reference laboratory team bi-monthly.

Given the large number of negative cases required and to avoid unnecessary delays to potential regulatory approval submissions, an interim review of the results by the data team and study investigators will be conducted when 172 positive cases have been recruited. The investigators will assess whether sufficient precision around the estimate for specificity has already been achieved for regulatory approval purposes and whether additional recruitment is required.

I. Ease-of-use questionnaire

At the beginning (following training) and at the end of the study, all the staff responsible for performing the RDTs will be asked to answer a short ease-of-use questionnaire. The questions will seek to capture the perceived ease of use of the RDT including the clarity of instructions for use and package labelling, the clinical sampling procedure, the reading time, the volume of specimen to be used, the ease/difficulty of the steps to perform the test (including sample preparation and application of the sample), the ease of reading and interpreting the results and perceived biosafety.

J. Data entry

Data will be collected using an electronic case report form (eCRF) form prior to sample collection and will match the data collected on the mandatory national surveillance paper form. Data will be entered into TERANGA Mobile, Institut Pasteur de Dakar's secure surveillance and clinical data collection system, on which the study team will be trained during study implementation. The study facilitator at each site will have responsibility to ensure that the eCRF is correctly completed and saved. In addition to the patient or caregiver interview, additional information may be supplemented through the national paper surveillance form or vaccination records (e.g. to obtain dates of vaccination).

K. Quality control (monitoring) and assurance (audit)

Quality control will be performed at each stage of data processing to ensure that all data are reliable and have been processed correctly. The study sites will be responsible for regularly checking the quality of the data they generates including whether all included patients have consent forms and have undergone all required sampling procedures.

IPD will conduct risk-based monitoring of the study and associated quality control checks as described in the detailed monitoring plan. Study monitors will review and verify source data to confirm that the data entered are accurate and complete and can be verified in the source documents; that the safety and rights of participants are protected; and that the study is being conducted in accordance with the current authorized protocol, Good Clinical Practice (GCP), and all applicable regulatory requirements. The monitoring plan will detail the frequency of monitoring visits and audits at the study site.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting at study sites:

* For whom confirmatory diagnostic testing is currently indicated as per the national surveillance protocol
* With clinical signs and symptoms consistent with the WHO suspected measles case definition including: History of fever, or observed fever (>37.5C) at presentation and a (non-vesicular) maculopapular rash; or clinically suspected measles
* ≤ 28 days after the onset of a rash
* Who if <18 years of age, have written, informed consent from their legal guardian (and verbally assent if more than 7 years old)
* Who if more than 18 years, give written, informed consent

Exclusion Criteria:

* Withdrawal of consent or assent as described above, at any time.
* Unsuccessful venous blood sampling after a maximum of 3 attempts, or a serum sample is no longer available for any reason.
* Clinical signs or symptoms requiring immediate referral/transfer of the patient to another site or centre, and/or for whom participation would involve a delay of urgent clinical interventions or investigations (i.e. potential inclusion of patients requiring immediate clinical management should be deferred until the patient is clinically stable).
* Clinical signs or symptoms that may be exacerbated by blood draw or upper respiratory sampling (e.g. stridor or severe respiratory distress)

Participants who meet the inclusion criteria should be included in the study but without oral fluid sampling if:

* They have a sore mouth or gums that would be exacerbated with oral fluid sampling
* They are significantly dehydrated and the mouth is very dry
* They refuse or are not able to cooperate with oral fluid sampling

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (all ages) presenting to participating health centres with signs and symptoms consistent with being a suspected measles case (WHO definition), for whom diagnostic testing is indicated for laboratory confirmation for national measles and rubella surveillance purposes in Senegal.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The clinical diagnostic performance of the RDT for measles case-confirmation using capillary blood by non-laboratory professional personnel under field conditions | 6 months
  Sensitivity and specificity of the RDT compared to the current laboratory reference standard using anti-measles IgM in serum by Enzyme Immuno Assay (EIA) and/or RT PCR of oral fluid, with 95% exact (Clopper Pearson) confidence intervals. The following stratified analyses will estimate the performance of the RDT by:
  * Site
  * Time since symptom onset (<7days; 7 to <14 days; ≥14 days)
  * Time since rash onset (<4 vs ≥days)
  * Age group (<1; 1 to <5; 5 to <16; 16+ years)
  * Recent vaccination status (in last 30 days and 60 days)
  * Rheumatoid factor status
  * RDT lots (if applicable)

SECONDARY OUTCOMES:
The clinical diagnostic performance of the RDT for measles case-confirmation using oral fluid by non-laboratory professional personnel under field conditions | 6 months
  Sensitivity and specificity of the RDT compared to the current laboratory reference standard using anti-measles IgM in serum by Enzyme Immuno Assay (EIA) and/or RT PCR of oral fluid, with 95% exact (Clopper Pearson) confidence intervals. The following stratified analyses will estimate the performance of the RDT by:
  * Site
  * Time since symptom onset (<7days; 7 to <14 days; ≥14 days)
  * Time since rash onset (<4 vs ≥days)
  * Age group (<1; 1 to <5; 5 to <16; 16+ years)
  * Recent vaccination status (in last 30 days and 60 days)
  * Rheumatoid factor status
  * RDT lots (if applicable)
The clinical diagnostic performance of the RDT for measles case-confirmation using serum by laboratory personnel | 6 months
  Sensitivity and specificity of the RDT compared to the current laboratory reference standard using anti-measles IgM in serum by Enzyme Immuno Assay (EIA) and/or RT PCR of oral fluid, with 95% exact (Clopper Pearson) confidence intervals. The following stratified analyses will estimate the performance of the RDT by:
  * Site
  * Time since symptom onset (<7days; 7 to <14 days; ≥14 days)
  * Time since rash onset (<4 vs ≥days)
  * Age group (<1; 1 to <5; 5 to <16; 16+ years)
  * Recent vaccination status (in last 30 days and 60 days)
  * Rheumatoid factor status
  * RDT lots (if applicable)
Inter-reader agreement by non-laboratory personnel of the RDT for measles case confirmation by IgM detection in capillary blood under field conditions | 6 months
  Results of inter-reader agreement will be displayed for each test on a 2x2 contingency table with, in each cell, the number of agreements/disagreements between the two readers. The concordance (of the qualitative interpretations of the RDT results) between the two readers will be evaluated using Cohen's kappa coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Cheikh Tidiane Diagne, PhD, Principal Investigator — Institut Pasteur de Dakar; Boly Diop, Principal Investigator — Ministry of Health, Senegal